CLINICAL TRIAL: NCT07218497
Title: Investigating the Evolutionary Impact of Metabolic Flexibility on Physical Activity-Dependent BDNF and Cognition: Insights From the Val66Met Polymorphism
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, David Raichlen, Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: APP-24-05903
Record Dates: First submitted 2025-09-12; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cognition; BDNF
Keywords: Cognition; BDNF; Val66Met SNP; Physical Activity; Ketosis
MeSH Terms: conditions — Motor Activity; Ketosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketosis Trial (Experimental): Participants will be given a sugar-free electrolyte mixture with d-beta-hydroxybutrate to drink in a 1:1 ratio calculated to 0.1816g/lb based on body weight before the treadmill test.
  Interventions: Drug: d-beta-hydroxybutrate
- Placebo Trial (Placebo Comparator): Participants consume a placebo consisting of a pure sugar-free electrolyte drink before treadmill test. The grams of placebo will be calculated 0.1816g/lb based on body weight.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: d-beta-hydroxybutrate — During the ketosis trial, participants will be given d-beta-hydroxybutrate mixed with sugar-free gatorade in a 1:1 ratio. This is to ensure the participant's electrolytes are high and to mask the bitter taste of d-beta-hydroxybutrate. The dosage per participant will be calculated 0.1816g/lb based on body weight to ensure participants remain in a state of ketosis for a minimum of 2 hours.
  Other Names: Ketosis Supplement
  Arms: Ketosis Trial
Drug: Placebo — Participants will consume a placebo consisting of a pure electrolyte drink.
  Arms: Placebo Trial

SUMMARY:
The goal of this clinical trial is to learn if a state of ketosis and physical activity will increase serum BDNF concentrations and improve cognition, specifically in individuals who possess the Met allele from the BDNF Val66Met SNP. The main questions it aims to answer are:

* Does the combination of ketosis and physical activity increase serum BDNF concentrations and cognition?
* Do Met Carriers of the BDNF Val66Met SNP demonstrate a significantly larger change in serum BDNF after physical activity and a state of ketosis compared to Val/Val Homozygotes?
* Do Met Carriers of the BDNF Val66Met SNP demonstrate a significantly larger increase in cognition after physical activity and a state of ketosis compared to Val/Val Homozygotes?

Researchers will compare a ketosis supplement to a placebo (a look-alike substance that contains no drug) to see if the ketosis supplement and physical activity increases serum BDNF and improves cognition.

Participants will:

* Participate in a drug trial where they will be given the ketosis supplement, and a placebo trial where they will ingest a placebo.
* Participants will donate a whole blood sample and take a cognitive test before and after the ketosis and placebo trial.
* Participants will take a 30-minute treadmill test during both the ketosis and placebo trial, after ingesting either the drug or placebo for each respective trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults
* 18 years old to 35 years old
* give informed consent

Exclusion Criteria:

* Diabetics
* history of low blood sugar
* limited physical abilities unable to participate in an aerobic treadmill test

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Serum BDNF | baseline, pre-intervention/procedure/surgery, and immediately after the intervention/procedure/surgery
  Whole blood will be taken from participants before and after the treadmill test for both placebo and ketosis trial days. Serum will be extracted and an ELIZA will be run to assess serum BDNF concentrations.

SECONDARY OUTCOMES:
Cognition | baseline, pre-intervention/procedure/surgery, and immediately after the intervention/procedure/surgery
  RBANS, Repeatable Battery for the Assessment of Neuropsychological Status, will be administered to participants before and after each respective trial day, both placebo and ketosis trials.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
At this time we do not intend to share IPD to protect their anonymity